CLINICAL TRIAL: NCT05488990
Title: Phase I, Single-center, Randomized, Controlled Trial to Evaluate the Antipsoriatic Efficacy of Calcipotriol in Novel Formulations Compared to Marketed Calcipotriol Products and Evaluation of Their Cutaneous Safety in a Psoriasis Plaque Test
Brief Title: Efficacy and Safety of Novel Formulations of Topical Calcipotriol in Patients With Mild to Moderate Plaque Psoriasis
Acronym: AKVANO-AKP01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lipidor AB (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALC01 / 310905BS; 2012-003951-12 (EudraCT Number)
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis plaque test; sonographic measurement; psoriatic infiltrate; clinical efficacy assessments; cutaneous safety; calcipotriene; calcipotriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm with several test fields (Experimental): Altogether six test fields (two active formulations, their corresponding vehicles and two comparators) located on the torso, or the extremities were randomly assigned for treatments per subject.
  Interventions: Drug: AKVANO-Calcipotriol formulation 1; Drug: AKVANO-Calcipotriol formulation 2; Drug: AKVANO vehicle formulation 1; Drug: AKVANO vehicle formulation 2; Drug: Daivonex solution; Drug: Daivonex cream

INTERVENTIONS:
Drug: AKVANO-Calcipotriol formulation 1 — Novel lipid based formulation (AKVANO) type 1 containing Calcipotriol (50 μg/g)
  Other Names: AKVC01
Drug: AKVANO-Calcipotriol formulation 2 — Novel lipid based formulation (AKVANO) type 2 containing Calcipotriol (50 μg/g)
  Other Names: AKVC02
Drug: AKVANO vehicle formulation 1 — Novel lipid based formulation (AKVANO) vehicle 1
  Other Names: AKVC01 vehicle
Drug: AKVANO vehicle formulation 2 — Novel lipid based formulation (AKVANO) vehicle 2
  Other Names: AKVC02 vehicle
Drug: Daivonex solution — Daivonex solution containing Calcipotriol (50 μg/g)
Drug: Daivonex cream — Daivonex cream containing Calcipotriol (50 μg/g)

SUMMARY:
This was a Phase I, single-center, randomized, controlled trial to evaluate the antipsoriatic efficacy of calcipotriol in novel formulations based on AKVANO technology as compared to marketed calcipotriol products (Daivonex® solution and cream) and to evaluate their cutaneous safety in a psoriasis plaque test

DETAILED DESCRIPTION:
This study was conducted to evaluate the efficacy and cutaneous safety of calcipotriol (50 μg/g) in novel formulations (AKVANO®) as compared to their corresponding vehicle formulations and marketed calcipotriol formulations (Daivonex®) in a psoriasis plaque test. In total, 24 subjects with chronic psoriasis vulgaris were enrolled in this single-centre, randomized, vehicle and comparator-controlled clinical trial and were treated under occlusion over a 12-day treatment period (10 applications). The anti-psoriatic effect was evaluated by sonographic measurement of the psoriatic infiltrate and investigators' clinical efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria had to be met for inclusion of a subject in the clinical trial:

* Subjects with psoriasis vulgaris in a chronic stable phase and mild or moderate plaque(s) with up to three plaque areas sufficient for six treatment fields
* The target lesion(s) should have been on the trunk or extremities (excluding palms/soles); psoriatic lesion on the knees were not used as a target lesion
* Plaques to be treated should have had a comparable psoriatic infiltrate thickness of at least 200 μm
* The physical examination of the skin had to be without disease findings unless the investigator considered an abnormality to be irrelevant to the outcome of the clinical trial
* Female volunteers of childbearing potential had to be either surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 % per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices [IUDs], sexual abstinence or had a vasectomized partner
* Written informed consent obtained

Exclusion Criteria:

Subjects were excluded from the clinical trial when one or more of the following conditions were met:

* Other skin disease noted on physical examination that was considered by the investigator to be relevant to the outcome of the trial;
* Subjects with psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, psoriasis arthropathica and pustular psoriasis
* Any topical antipsoriatic treatment on the plaques to be treated in this trial (including corticosteroids, except for salicylic acid) in the three months before first treatment and/or during the trial
* Systemic treatment with antipsoriatics e.g. corticosteroids, cytostatics, retinoids in the three months before first treatment and during the trial
* Treatment with systemic or locally acting medications which might have countered or influenced the trial aim (medications which were known to provoke or aggravate psoriasis, e.g. ß-blocker, antimalarial drugs, lithium) within three months before first treatment and/or during the trial
* Known allergic reactions irritations or sensitivity to the active ingredients or other components of the investigational products;
* Contraindications according to summary of product characteristics of Daivonex®
* Evidence of drug or alcohol abuse
* Pregnancy or nursing
* UV-therapy within four weeks before first treatment and during the trial
* Symptoms of a clinically significant illness that might have influenced the outcome of the trial in the four weeks before first treatment and during the trial
* Participation in the treatment phase of another clinical trial within the last four weeks prior to the first treatment in this clinical trial
* In the opinion of the investigator or physician performing the initial examination the subject should not have participated in the clinical trial, e.g. due to probable non-compliance or inability to understand the trial and give adequately informed consent
* Close affiliation with the investigator (e.g. a close relative) or persons working at bioskin GmbH or subject was an employee of sponsor
* Subject was institutionalized because of legal or regulatory order

Ages: 32 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2013-06-17 (Actual); Study Completion 2013-06-17 (Actual)

PRIMARY OUTCOMES:
Comparison of AKVANO-Calcipotriol formulations to their corresponding vehicles in terms of change in infiltrate thickness from baseline to Day 12 | 12 days
  The thickness of psoriatic infiltrate will be recorded as echo lucent psoriatic band (ELB) using a 20 MHz high frequency sonograph (PROFI USB, Taberna pro Medicum, Lueneburg) on day 1 (baseline) and day 12 (end of treatment; EoT). Mean change of infiltrate thickness will be determined.

SECONDARY OUTCOMES:
Comparison of AKVANO-Calcipotriol formulations to their corresponding comparators (Daivonex solution and cream) in terms of change in infiltrate thickness from baseline to Day 12 | 12 days
  The thickness of psoriatic infiltrate will be recorded as echo lucent psoriatic band (ELB) using a 20 MHz high frequency sonograph (PROFI USB, Taberna pro Medicum, Lueneburg) on day 1 (baseline) and day 12 (end of treatment; EoT). Mean change of infiltrate thickness will be determined.
Comparison of AKVANO-Calcipotriol formulations to their corresponding vehicles and comparators in terms of change in infiltrate thickness and Area under curve (AUC) of change in infiltrate thickness from baseline to Day 8 | 8 days
  The thickness of psoriatic infiltrate will be recorded as echo lucent psoriatic band (ELB) using a 20 MHz high frequency sonograph (PROFI USB, Taberna pro Medicum, Lueneburg) on day 1 (baseline) and day 8. Mean change of infiltrate thickness and AUC of infiltrate thickness will be determined.
Clinical assessment of the treatment efficacy of all formulations at day 8 | 8 days
  Clinical assessment (global assessment) of the test fields will be made at visit (day 8 and 12) after day 1 using a defined five-point scale of worsened (-1), unchanged (0), slight improvement (1), clear improvement but not completely healed (2) and completely healed (3). The comparison of single test fields will be made to the untreated plaque(s) beneath the hydrocolloid dressing and next to the respective test field. Clinically apparent differences in erythema and infiltration will contribute to this global assessment. At baseline (Day 1) the score will be documented as "0" (unchanged).
Clinical assessment of the treatment efficacy of all formulations at day 12 | 12 days
  Clinical assessment (global assessment) of the test fields will be made at visit (day 8 and 12) after day 1 using a defined five-point scale of worsened (-1), unchanged (0), slight improvement (1), clear improvement but not completely healed (2) and completely healed (3). The comparison of single test fields will be made to the untreated plaque(s) beneath the hydrocolloid dressing and next to the respective test field. Clinically apparent differences in erythema and infiltration will contribute to this global assessment. At baseline (Day 1) the score will be documented as "0" (unchanged).

OTHER OUTCOMES:
All Adverse events (AEs) (non-treatment-emergent and treatment-emergent) will be documented. | 12 days
  All Adverse events (AEs) (non-treatment-emergent and treatment-emergent) will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Siemetzki, MD, Principal Investigator — Bioskin GmbH
Locations (1):
- bioskin GmbH, Bergmannstrasse, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmback J, Rinwa V, Halthur T, Rinwa P, Carlsson A, Herslof B. AKVANO(R): A Novel Lipid Formulation System for Topical Drug Delivery-In Vitro Studies. Pharmaceutics. 2022 Apr 5;14(4):794. doi: 10.3390/pharmaceutics14040794. PMID 35456628